CLINICAL TRIAL: NCT03909893
Title: A Study of Adaptive Radiation Therapy for Pelvic Genitourinary Cancer
Acronym: ARTGU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is being closed. The protocol may be reviewed and consolidated under a new study currently in development.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5929
Record Dates: First submitted 2018-05-14; First posted 2019-04-10 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Bladder Cancer
Keywords: Adaptive; Radiation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Radiation Therapy (Experimental)
  Interventions: Radiation: Adaptive Radiation Therapy

INTERVENTIONS:
Radiation: Adaptive Radiation Therapy — Cone-beam CT images as well as MRI scans will be used to make any changes to the radiation treatment plan, part of the way through the treatment. Adaptation of treatment plans may allow smaller target volumes to be treated with higher doses, while minimizing the side effects to surrounding organs.

SUMMARY:
Radical radiation therapy for prostate cancer is a common treatment that has shown to improve clinical outcomes in a post-operative setting. However, radiation therapy after surgery poses a greater risk for bladder and rectum injury for patients with prostate or bladder cancer. For prostate cancer patients, the risk is further amplified when pelvic nodes are part of the target irradiated volume. For bladder cancer patients, the risk of injury increases when more of the bladder is part of the target volume. Using an adaptive radiation therapy approach allows for correcting any shifts in the target volume. ART approach uses images from treatment to adapt the treatment plan. This study will use Adaptive Radiation Therapy for patients who receive pelvic nodal radiotherapy for either prostate or bladder cancer. Their treatment plans will adapted using MRI scans and CBCT scans taken during their first week of radiotherapy to account for any shifts in the target volume. The purpose of this study is to evaluate the feasibility of ART approach and its and on treatment plan quality metrics for pelvic radiotherapy. Acute and late toxicities will also be evaluated. 40 participants (minimum of 10 bladder cancer patients) will be enrolled. The participants will be followed for a period of 5 years post radiation therapy, during which they will have PSA as per standard practice, along with follow-up questionnaires (EPIC for prostate cancer patients and BUSS for bladder cancer patients).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of adenocarcinoma of the prostate after radical prostatectomy:

   * Clinical stage pT3, pT4, or pT2 with positive margin; OR,
   * any p-stage with persistently elevated post-operative PSA > 0.05ng/mL; OR,
   * a delayed rise in PSA post-operative
2. Histologic diagnosis of transitional cell carcinoma of the bladder with intact bladder and:

   * Clinical stage cT2, cT3, cT4, and N0 or N1

Exclusion Criteria:

1. Inflammatory bowel disease or other contraindications to radiotherapy.
2. Prior pelvic radiotherapy
3. Previous cytotoxic chemotherapy
4. Evidence of systemic metastases on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Dosimetry | 5 years
  Difference in dose-volume irradiation of critical organs between original and adapted plan will be compared.

SECONDARY OUTCOMES:
Toxicity in Patients | Before Radiation Therapy, and at Month 3, Year 1, 3 & 5 after Radiation Therapy
  To determine a preliminary measure of toxicity with this technique. CTCAE toxicity data will be described for this population.
Bladder Cancer Patients' Quality of Life Function | Before Radiation Therapy, and at Month 3, Year 1, 3 & 5 after Radiation Therapy
  Bladder Utility Symptom Scale (BUSS) questionnaires will be scored and analyzed to determine QoL function. BUSS will be scored (1-100) as per standard criteria. Data will be analyzed as a continuous variable
Prostate Cancer Patients' Quality of Life Function | Before Radiation Therapy, and at Month 3, Year 1, 3 & 5 after Radiation Therapy
  Expanded Prostate Cancer Index Composite (EPIC) questionnaires will be scored and analyzed to determine QoL function. EPIC will be scored (1-100) as per standard criteria. Data will be analyzed as a continuous variable
Biochemical Control in Prostate Patients | PSA will be done before Radiation Therapy, and at Month 3, Year 1, 3 and 5 after Radiation Therapy
  For prostate patients, patients will be considered to have biochemical failure if the PSA has risen 2ng above nadir.
Local Control in Bladder Patients | 5 years
  Local control will be defined by an absence of clinically locally recurrent disease
Feasibility of the use of Fiducial markers for bladder RT: quality of target delineation using fiducial markers | 5 years
  Feasibility will be determined by analyzing the quality of target delineation using fiducial markers in bladder cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MD, Principal Investigator — Princess Margaret Cancer Centre - University Health Network
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada